CLINICAL TRIAL: NCT00751621
Title: A Multicenter Extension Study of the Efficacy, Tolerability, and Safety of Immune Globulin Subcutaneous (Human) IgPro20 in Subjects With Primary Immunodeficiency (IgPro20 EU Extension Study)
Brief Title: Study of Subcutaneous Immune Globulin in Patients Requiring IgG Replacement Therapy (EU Extension Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLB07_002CR; 1472 (Other: CSL Behring); 2008-000830-30 (EudraCT Number)
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2012-12

CONDITIONS: Primary Immunodeficiency (PID)
Keywords: Immune globulin subcutaneous; SCIG; primary immunodeficiency; PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Hizentra; Immunoglobulin G; Proline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IgPro20 (Experimental): Subcutaneous (SC) administration by the subject/parent/guardian with the planned weekly dose of IgPro20 to be the same as the subject's last dose recommended by the investigator in study ZLB06_001CR (NCT00542997).
  Interventions: Biological: IgPro20

INTERVENTIONS:
Biological: IgPro20
  Other Names: IgG with Proline (IgPro); Hizentra

SUMMARY:
This study is a continuation of the study ZLB06_001CR with the objective of assessing efficacy, tolerability, safety of IgPro, as well as long-term health-related quality of life in patients with PID.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with primary humoral immunodeficiency, namely with a diagnosis of Common variable immunodeficiency (CVID) as defined by the Pan-American Group for Immunodeficiency (PAGID) and the European Society for Immunodeficiencies (ESID), or X-linked agammaglobulinemia (XLA) as defined by PAGID and ESID, or autosomal recessive agammaglobulinemia who have participated in the study ZLB06_001CR and who have tolerated IgPro well
* Written informed consent

Exclusion Criteria:

* Hypoalbuminemia, protein-losing enteropathies, and any proteinuria (defined as total urine protein concentration > 0.2g/L)
* Other significant medical conditions that could increase the risk to the subject
* Females who are pregnant, breast feeding or planning a pregnancy during the course of the study
* Participation in a study with an investigational medicinal product within three months prior to enrollment, except for ZLB06_001CR
* Evidence of uncooperative attitude
* Any condition that is likely to interfere with evaluation of the IMP or satisfactory conduct of the study
* Subjects who are employees at the investigational site, relatives or spouse of the investigator

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (13):
- Study Site, Paris, France
- Germany (4):
  - Study Site, Berlin
  - Study Site, Freiburg im Breisgau
  - Study Site, Leipzig
  - Study Site, Mainz
- Study Site, Warsaw, Poland
- Romania (2):
  - Study Site, Cluj-Napoca
  - Study Site, Timișoara
- Spain (2):
  - Study Site, Barcelona
  - Study Site, Seville
- Study Site, Gothenburg, Sweden
- Study Site, Bern, Switzerland
- Study Site, London, United Kingdom

REFERENCES:
- [Result] Jolles S, Borte M, Nelson RP Jr, Rojavin M, Bexon M, Lawo JP, Wasserman RL. Long-term efficacy, safety, and tolerability of Hizentra(R) for treatment of primary immunodeficiency disease. Clin Immunol. 2014 Feb;150(2):161-9. doi: 10.1016/j.clim.2013.10.008. Epub 2013 Oct 26. PMID 24412910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who had previously participated in the pivotal study ZLB06_001CR (NCT00542997) were enrolled in the extension study ZLB07_002CR.
Period: Overall Study
Arm/Group | IgPro20
Started | 40
Completed | 36
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Subject moved to another country | 1
Not completed — Poor adherence to asthma treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | IgPro20
Number analyzed (Participants) | 40
Age, Customized [Number; unit: participants]
  2 to < 12 years | 15
  12 to < 16 years | 4
  16 to < 65 years | 21
  ≥ 65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Total Serum IgG Trough Levels
Description: The IgG trough values per subject were aggregated to a median value, and then median values across subjects were summarized using descriptive statistics.
Time Frame: Up to 42 months
Population: The "all treated" (AT) safety data set comprised all subjects treated with IgPro20 during any study period and was identical to the "Full Analysis/intention-to-treat" (ITT) data set that comprised all subjects treated with IgPro20 and for whom any efficacy data was available.
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- IgPro20: Subcutaneous administration by the subject/parent/guardian with the planned weekly dose of IgPro20 to be the same as the subject's last dose recommended by the investigator in study ZLB06_001CR (NCT00542997).
Arm/Group | IgPro20
Number analyzed (Participants) | 40
g/L | 7.97 (1.171)

2. Secondary Outcome: Annualized Rate of Clinically Documented Serious Bacterial Infections (SBIs)
Description: The annualized rate was based on the total number of SBIs and the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
  Potential SBIs included bacterial pneumonia, bacteremia and septicemia, osteomyelitis/septic arthritis, bacterial meningitis, and visceral abscess. If an adverse event (AE) was identified as a potential SBI, the AE was adjudicated by the Medical Monitor and Investigator to determine if the event fulfilled the predefined criteria for SBIs.
Time Frame: Up to 42 months
Population: The AT safety data set comprised all subjects treated with IgPro20 during any study period and was identical to the ITT data set that comprised all subjects treated with IgPro20 and for whom any efficacy data was available.
Measure: Number; unit: SBIs per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 40
Number analyzed (Subject Study Days) | 38208
SBIs per subject year
  Annualized Rate | 0.048
  Upper 1-sided 99% Confidence Limit | 0.1252

3. Secondary Outcome: Annualized Rate of Infection Episodes
Description: The annualized rate was based on the total number of infection episodes occurring during the study divided by the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
Time Frame: Up to 42 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: infection episodes per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 40
Number analyzed (Subject Study Days) | 38208
infection episodes per subject year | 3.334 [2.993 to 3.703]

4. Secondary Outcome: Number of Infection Episodes
Description: Total number of infections for the specified analysis population
Time Frame: Up to 42 months
Population: as for outcome 2
Measure: Number; unit: infection episodes
Arm/Group | IgPro20
Number analyzed (Participants) | 40
infection episodes | 349

5. Secondary Outcome: Annualized Rate of Days Out of Work / School / Kindergarten / Day Care or Unable to Perform Normal Activities Due to Infections
Description: The annualized rate was based on the total number of days out of work / school / kindergarten / day care or inability to perform normal activities due to infection, and the total number of subject diary days for all subjects in the specified analysis population and adjusted to 365 days.
Time Frame: Up to 42 months
Population: as for outcome 2
Measure: Number; unit: days per subject year
Units Other Than Participants: Subject Diary Days
Arm/Group | IgPro20
Number analyzed (Participants) | 40
Number analyzed (Subject Diary Days) | 38045
days per subject year | 6.773

6. Secondary Outcome: Number of Days Out of Work / School / Kindergarten / Day Care or Unable to Perform Normal Activities Due to Infections
Description: Total number of days out of work / school / kindergarten / day care or unable to perform normal activities due to infections, for the specified analysis population
Time Frame: Up to 42 months
Population: as for outcome 2
Measure: Number; unit: days
Arm/Group | IgPro20
Number analyzed (Participants) | 40
days | 706

7. Secondary Outcome: Annualized Rate of Hospitalization Due to Infections
Description: The annualized rate was based on the total number of days of hospitalization due to infections and the total number of subject diary days for all subjects in the specified analysis population and adjusted to 365 days.
Time Frame: Up to 42 months
Population: as for outcome 2
Measure: Number; unit: days per subject year
Units Other Than Participants: Subject Diary Days
Arm/Group | IgPro20
Number analyzed (Participants) | 40
Number analyzed (Subject Diary Days) | 38045
days per subject year | 1.055

8. Secondary Outcome: Number of Days of Hospitalization Due to Infections
Description: Total number of days of hospitalization due to infections for the specified analysis population
Time Frame: Up to 42 months
Population: as for outcome 2
Measure: Number; unit: days
Arm/Group | IgPro20
Number analyzed (Participants) | 40
days | 110

9. Secondary Outcome: Use of Antibiotics for Infection Prophylaxis and Treatment
Description: Annualized rate of days with antibiotics for infection prophylaxis and treatment. The annualized rate was based on the total number of days of antibiotic use for infection prophylaxis and treatment in the efficacy period, and the total number of subject study days for all subjects in the specified analysis population, and adjusted to 365 days.
Time Frame: Up to 42 months
Population: as for outcome 2
Measure: Number; unit: days per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 40
Number analyzed (Subject Study Days) | 38208
days per subject year | 72.13

10. Secondary Outcome: Health Related Quality of Life (Short Form 36 Health Survey)
Description: The Short Form 36 Health Survey (SF-36) is a 36-item questionnaire that measures generic health concepts that are relevant across age, disease, and treatment groups. The questions are grouped into eight domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 100, with higher scores indicating a better health state.
Time Frame: At baseline and at the last available post-baseline observation for each subject (up to 42 months)
Population: The analysis population comprised the Full-Analysis health related quality of life (HRQL) data set (defined as all subjects entered into the study who complete a baseline and at least 1 follow-up HRQL assessment), who were at least 15 years of age.
Measure: Median (Full Range); unit: score on a scale
Groups:
- IgPro20 - At Baseline: SF-36 score at baseline.
- IgPro20 - At End of Study: SF-36 score at end of study (defined as the last available post-baseline observation for each subject).
Arm/Group | IgPro20 - At Baseline | IgPro20 - At End of Study
Number analyzed (Participants) | 20 | 20
score on a scale
  Physical Functioning | 95.0 [75.0 to 100.0] | 100.0 [20.0 to 100.0]
  Role-physical | 100.0 [18.8 to 100.0] | 100.0 [37.5 to 100.0]
  Role-emotional | 100.0 [25.0 to 100.0] | 100.0 [25.0 to 100.0]
  Social Functioning | 100.0 [62.5 to 100.0] | 100.0 [37.5 to 100.0]
  Bodily Pain | 84.0 [22.0 to 100.0] | 84.0 [22.0 to 100.0]
  Mental Health | 85.0 [55.0 to 95.0] | 80.0 [35.0 to 95.0]
  Vitality | 65.6 [31.3 to 81.3] | 75.0 [18.8 to 100.0]
  General Health | 52.0 [15.0 to 82.0] | 54.5 [20.0 to 92.0]

11. Secondary Outcome: Clinically Relevant Changes in Vital Signs From Baseline to the Completion Visit.
Description: The total number of subjects with clinically relevant changes in vital signs from baseline to the completion visit. Vital signs included heart rate, systolic blood pressure, diastolic blood pressure, and body temperature.
Time Frame: At baseline (data either from Infusion 40 or the completion visit of study ZLB06_001CR), and at completion (up to 42 months).
Population: The AT safety data set (which comprised all subjects treated with IgPro20 during any study period and was identical to the ITT data set that comprised all subjects treated with IgPro20 and for whom any efficacy data was available) and for whom vital signs data was collected at both baseline and completion.
Measure: Number; unit: participants
Arm/Group | IgPro20
Number analyzed (Participants) | 39
participants | 0

12. Secondary Outcome: Clinically Significant Abnormal Changes in Routine Laboratory Parameters Between Baseline and the Completion Visit.
Description: The total number of subjects with clinically significant abnormal changes in routine laboratory parameters between baseline and the completion visit. Routine laboratory parameters included haematology, serum chemistry and urinalysis.
Time Frame: as for outcome 11
Population: The AT safety data set (which comprised all subjects treated with IgPro20 during any study period and was identical to the ITT data set that comprised all subjects treated with IgPro20 and for whom any efficacy data was available) and for whom laboratory parameter data was collected at both baseline and completion.
Measure: Number; unit: participants
Arm/Group | IgPro20
Number analyzed (Participants) | 40
participants
  Haematology | 3
  Serum Chemistry | 1
  Urinalysis | 0

13. Secondary Outcome: Rate, Severity and Relatedness of Any Adverse Events (AEs) Per Infusion
Description: The rate of AEs was the number of AEs over the number of infusions administered. Mild AE: Did not interfere with routine activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities. At least possibly related AEs included possibly related AEs, probably related AEs, and related AEs.
Time Frame: Up to 42 months
Population: The AT safety data set comprised all subjects treated with IgPro20 during any study period.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Number of Infusions
Arm/Group | IgPro20
Number analyzed (Participants) | 40
Number analyzed (Number of Infusions) | 5405
AEs per infusion
  Total AEs | 0.0936
  Mild AEs | 0.0685
  Moderate AEs | 0.0231
  Severe AEs | 0.0020
  At least possibly related AEs | 0.0026
  Serious AEs | 0.0033
  At least possibly related and serious AEs | 0

ADVERSE EVENTS:
Time Frame: AEs were collected for the duration of the study, up to 42 months.
Description: A total of 5405 weekly infusions of IgPro20 were administered to 40 subjects in this study. Three subjects received fewer than 100 infusions. The AT safety data set comprised all subjects treated with IgPro20 during any study period. AEs in "General disorders" were collected under the MedDRA SOC General disorders and administration site conditions.
Arm/Group | IgPro20
Serious Adverse Events (participants affected / at risk) | 14/40
Other Adverse Events (participants affected / at risk) | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=40)
Pneumonia bacterial (Infections and infestations) | 5 (5)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1)
Face oedema (General disorders) | 1 (1) — This AE was collected under the MedDRA System Organ Class (SOC) General disorders and administration site conditions.
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=40)
Bronchitis (Infections and infestations) | 21 (51)
Upper respiratory tract infection (Infections and infestations) | 18 (49)
Sinusitis (Infections and infestations) | 13 (31)
Nasopharyngitis (Infections and infestations) | 12 (19)
Rhinitis (Infections and infestations) | 9 (15)
Febrile infection (Infections and infestations) | 6 (10)
Acute sinusitis (Infections and infestations) | 5 (5)
Pharyngitis (Infections and infestations) | 5 (10)
Influenza (Infections and infestations) | 4 (4)
Viral infection (Infections and infestations) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 4 (5)
Conjunctivitis infective (Infections and infestations) | 3 (11)
Ear infection (Infections and infestations) | 3 (6)
Enteritis infectious (Infections and infestations) | 3 (12)
Lower respiratory tract infection (Infections and infestations) | 3 (6)
Oral herpes (Infections and infestations) | 3 (8)
Otitis media (Infections and infestations) | 3 (8)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (6)
Acute tonsillitis (Infections and infestations) | 2 (3)
Diarrhoea infectious (Infections and infestations) | 2 (3)
Enterobiasis (Infections and infestations) | 2 (3)
Gastroenteritis (Infections and infestations) | 2 (2)
Laryngitis (Infections and infestations) | 2 (6)
Otitis externa (Infections and infestations) | 2 (2)
Otitis media acute (Infections and infestations) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (34)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (9)
Diarrhoea (Gastrointestinal disorders) | 3 (5)
Aphthous stomatitis (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Pyrexia (General disorders) | 4 (6)
Chest pain (General disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Dizziness (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 2 (6)
Sciatica (Nervous system disorders) | 2 (2)
Weight increased (Investigations) | 3 (5)
Wisdom teeth removal (Surgical and medical procedures) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.